CLINICAL TRIAL: NCT04783987
Title: Gait Parameters Under Single and Dual Task Conditions in Children With Specific Learning Difficulties: A Case-control Study
Brief Title: Single and Dual Task Gait Parameters in Children With Specific Learning Difficulties
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2020/333
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Specific Learning Disorder; Gait
MeSH Terms: conditions — Specific Learning Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control Group: Walking Assessments will be practised under dual and single task conditions.
  Interventions: Other: Walking asessments
- Case Group: Walking Assessments will be practised under dual and single task conditions.
  Interventions: Other: Walking asessments

INTERVENTIONS:
Other: Walking asessments — Gait parameters will be evaluated in single and dual task conditions with 10 Meter Walk Test and wireless digital miniature portable walking and movement analyzer.
  Other Names: 10 meter walking Test

SUMMARY:
Children with spesific learning disorders have differences in motor and cognitive abilities compared to normal developing children.

Motor tasks as walking are not just have a motor components and also require a cognitive process to realize. Therefore cognitive abilities may effect motor performance.

In daily life, individuals perform dual or multitasks instead of single tasks naturally. Dual task is defined as the concurrent performance of two tasks that can be performed independently. Also dual tasks may be created from different tasks combinations such as a motor-motor dual task or motor-cognitive dual task.

Therefore, aim of the study is to compare gait parameters with healthy controls in single and dual task conditions in children with Special Learning Difficulties.

DETAILED DESCRIPTION:
The fifth edition of the The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) opted for a categorical approach that introduced the Specific Learning Difficulties. Accordingly, it is thought that specific learning difficulties include many characteristics such as genetic risk, environmental risk factors, developmental characteristics, comorbidity and cognitive weaknesses. According to DSM-5, Specific Learning Difficulties are difficulties in using learning and school skills, which last at least six months, and are characterized by the presence of at least one of the following symptoms, despite the necessary attempts:

1. Slowness and mistakes in reading words
2. Difficulties in reading comprehension
3. Problems with spelling
4. Written expression difficulties
5. Number perception and calculation problems experienced
6. Numerical reasoning problems. In the literature, there are explanations about many cognitive limitations in children with specific learning difficulties, such as information processing, perceptual motor skills, processing of visual stimuli, phonological approach and the theory of cerebellum disorder. All of these cognitive limitations can also affect the dual task performance of these children.

In daily life, individuals perform dual or multitasks instead of single tasks naturally. Dual task is defined as the concurrent performance of two tasks that can be performed independently. Also dual tasks may be created from different tasks combinations such as a motor-motor dual task or motor-cognitive dual task.

However, no study investigating the effect of specific learning difficulties on walking parameters in single and dual task conditions has been found. In the light of the information is obtained from the literature, the gait parameters of children diagnosed with specific learning difficulties in single and dual task conditions may differ from the healthy control group. Therefore, this study's primary goal is to compare gait parameters in single and dual task conditions in children with Special Learning Disabilities with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Case Group

* To be in the age range of 6-17
* To have a diagnosis of special learning disability Control Group
* To be in the age range of 6-17
* To be physically, mentally and psychologically healthy

Exclusion Criteria:

* Any acute or chronic orthopedic or neurological disease that may affect walking performance,
* Any surgery within the last 6 months,
* A hearing impairment that cannot be corrected with a hearing aid
* A visual impairment that cannot be corrected with glasses.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: The case group of children between the ages of 6-17 who has been diagnosed with Specific Learning Difficulty and who attends the Specific Learning Difficulty Support Education Program of the Ministry of National Education regularly twice a week; It is planned that a healthy children between the ages of 6-17 will form the control group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Gait speed | 15 minutes
  The time it takes to walk a specified distance
Cadance | 15 minutes
  number of steps per minute
Strength length | 15 minutes
  It is the distance between points where the same heel touches the ground twice in a row.

CONTACTS AND LOCATIONS:
Overall Officials: Emel TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)